CLINICAL TRIAL: NCT07019324
Title: Evaluation of Cognitive Disorders and Serum BDNF/ProBDNF Levels in Cancer Patients Receiving Chemotherapy
Brief Title: BDNF Levels in Cancer Patients Receiving Chemotherapy
Acronym: CARE
Status: Active, not recruiting | Type: Observational
Sponsor: Cemre Aydeğer (Other)
Responsible Party: Sponsor-Investigator, Cemre Aydeğer, Çanakkale Onsekiz Mart University, Çanakkale Onsekiz Mart University
Organization: Çanakkale Onsekiz Mart University (Other)
Other Study IDs: TKB-2025-5052; TKB-2025-5052 (Other Grant/Funding Number: Çanakkale Onsekiz Mart University)
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-01

CONDITIONS: BDNF; Cognitive Functions; Chemotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Cognitive impairment following chemotherapy is defined as chemotherapy-induced cognitive impairment (CCIID). CCIID, which significantly reduces the quality of life of cancer patients receiving chemotherapy, develops as a result of neurotoxicity. It is stated that 75% of patients receiving chemotherapy have cognitive changes. In addition, 35% of patients complain of various cognitive impairments (hearing, perception, decision-making, etc.) for a few months after chemotherapy ends. This situation makes life conditions very difficult for patients who are already experiencing a very difficult disease and treatment process.

Brain-Derived Neurotrophic Factor (BDNF) is an extracellular signaling protein known for its dominant role in the development of the nervous system, such as neurogenesis, neuroprotection, neurodegeneration, synaptic plasticity, and resistance to neuronal stress. This protein has opposing effects with its mature form, pro-BDNF protein, and pro-BDNF/BDNF ratios affect neuronal health. Although a number of factors have been identified that are responsible for the deterioration of the cognitive levels of patients receiving chemotherapy, the role of BDNF and pro-BDNF levels in cognitive functions in cancer patients receiving chemotherapy is unknown. In light of this information, the aim of our study is to reveal the effects of chemotherapy-induced cognitive impairment (CIID) on pro-BDNF/BDNF levels and to evaluate the cognitive effects. In line with this aim, patients who apply to Çanakkale Onsekiz Mart University, Faculty of Medicine, Department of Oncology, Polyclinic and Chemotherapy Unit and who have not yet received their first chemotherapy will be included in the study. Before the first chemotherapy, during routine follow-ups in the 3rd month of chemotherapy and in the 6th month in Aydın, 1 extra tube of blood will be taken and BDNF levels will be examined. At the same time, the Montreal Cognitive Assessment (MoCA) test will be applied to the patients to evaluate their cognitive functions. Thus, serum BNDF, proBDNF levels will be determined and the BDNF/proBDNF ratio will be revealed.

DETAILED DESCRIPTION:
Detection of chemotherapy-induced cognitive impairment

ELIGIBILITY:
Inclusion Criteria:

* Cancer definations and decided the chemotherapy treatment

Exclusion Criteria:

* Having other disease whixh effected cognitive function
* Brain cancers
* Brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Applying Çanakkale Onsekiz Mart University Oncology Department
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-06-04 (Estimated); Study Completion 2026-06-04 (Estimated)

PRIMARY OUTCOMES:
BDNF level | Until 9 month
  BDNF level from every 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Çanakkale Onsekiz Mart University, Çanakkale, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided